CLINICAL TRIAL: NCT04462692
Title: A Prospective, Observational Study to Evaluate Ocular Disease Progression in Children With CLN2 Batten Disease
Brief Title: An Observational Study in Children With CLN2 Batten Disease
Status: Withdrawn | Type: Observational
Why Stopped: study stopped due to company decision
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGX-381-9101
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Neuronal Ceroid Lipofuscinosis Type 2 (CLN2)
Keywords: CLN2, Batten Disease
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, longitudinal natural history study to document the progression of ocular manifestations of CLN2 disease among a community-dwelling population of pediatric participants affected by this disease.

DETAILED DESCRIPTION:
CLN2 is a rare disease with limited available ocular natural history data. While current standard of care slows motor degeneration, it is not known to treat the ocular manifestations of disease. This study is planned to document, through prospective data collection, ocular disease progression in children with a clinical presentation consistent with CLN2 Batten disease undergoing current standard of care for their condition. No investigational product is administered in this observational study.

ELIGIBILITY:
Inclusion Criteria:

A participant is eligible to be included in the study only if all of the following criteria apply:

1. His or her legal guardian(s) is(are) willing and able to provide them written, signed informed consent.
2. Has documented diagnosis of CLN2 disease due to TPP1 deficiency, or has a relative clinically diagnosed with CLN2 with the same mutation as the participant
3. Is currently receiving biweekly ERT treatment with cerliponase alfa

Exclusion Criteria:

A participant is excluded from the study if any of the following criteria apply:

1. Has had prior treatment with an adeno-associated virus-based AAV gene therapy
2. Is currently participating in a clinical trial of investigational product for the treatment of CLN2 disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with CLN2 Batten disease undergoing current standard of care for their condition.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-03-31 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in retinal structure in children with CLN2 Batten disease | 96 weeks
  As assessed by SD-OCT measures over time.

SECONDARY OUTCOMES:
Change in visual function | 96 weeks
  As assessed by visual acuity over time.
Change in visual function | 96 weeks
  As assessed by pupillary light reflex over time.

IPD SHARING:
Plan to Share IPD: No